CLINICAL TRIAL: NCT05826197
Title: A Study on the Construction of a Comprehensive Predictive Model for Axillary Lymph Node Metastasis in Breast Cancer
Brief Title: Prediction of Axillary Lymph Node Metastasis Status in Breast Cancer Based on PET/CT Radiomics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-YBSF-480
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Axillary lymph node metastasis
  Interventions: Other: Radiomics
- No axillary lymph node metastasis

INTERVENTIONS:
Other: Radiomics — PET Radiomics
  Groups: Axillary lymph node metastasis

SUMMARY:
Patients with suspected breast cancer undergoing PET/CT at our hospital. The PET/CT center's chief physician and senior attending physician reviewed the films together and disagreement, if any, was resolved by consensus. The lesion was visually identified. A 3D region of interest(ROI) of the lesion was automatically outlined using the 40% threshold method, and PET metabolic parameters were measured . Breast lesions with radionuclide concentrations greater than those in normal breast tissue are considered to be breast cancer lesions, while lymph nodes with radionuclide concentrations greater than those in muscle tissue are considered to be metastatic lymph nodes.

Image segmentation: Image segmentation was performed using ITK-SNAP software (4) (version 3.6.0, http://www.itksnap.org/), Brush Style: circular, Brush Size: 10, Brush Options: 3D. The entire tumor volume was outlined on the PET image as ROI for segmentation.

An open source Python package (PyRadiomics version 3.0.1(5)) was used to extract the radiomics features from the ROI.

Univariate and multivariate binary logistic regressions were used to construct model for predicting lymph node metastasis in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1) 18F-FDG PET/CT for breast occupancy; 2) adult female patients with pathologically confirmed breast cancer (age ≥18 years); 3) no history of surgery, radiotherapy, or chemotherapy before 18F-FDG PET/CT; and 4) interval between 18F-FDG PET/CT and puncture/surgery ≤2 weeks.

Exclusion Criteria:

* 1) multifocal, bilateral, or occult breast cancer; 2) incomplete clinical or pathological data; 3) poor PET/CT image quality, when metabolic tumor volume(MTV) cannot be automatically segmented; and 4) concomitant malignant tumors.

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with breast cancer undergoing PET/CT at our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-10 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Radiomics score | 1 day During the inspection
  Higher radiomics scores indicate better model prediction performance

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li Y, Han D, Shen C. Prediction of the axillary lymph-node metastatic burden of breast cancer by 18F-FDG PET/CT-based radiomics. BMC Cancer. 2024 Jun 7;24(1):704. doi: 10.1186/s12885-024-12476-3. PMID 38849770
- [Derived] Li Y, Han D, Shen C, Duan X. Construction of a comprehensive predictive model for axillary lymph node metastasis in breast cancer: a retrospective study. BMC Cancer. 2023 Oct 24;23(1):1028. doi: 10.1186/s12885-023-11498-7. PMID 37875818